CLINICAL TRIAL: NCT01002534
Title: Does a Nasal Instillation of Vardenafil Normalize the Nasal Potential Difference in Cystic Fibrosis Patients Homozygous for the F508del Mutation? A Randomized, Double Blind, Placebo-controlled Study.
Brief Title: Does a Nasal Instillation of Vardenafil Normalize the Nasal Potential Difference in Cystic Fibrosis Patients?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not yet started
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VARD-99
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Vardenafil; Nasal instillation; Nasal Potential difference
MeSH Terms: conditions — Cystic Fibrosis | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- baseline (No Intervention): visit 1
- Vardenafil (Active Comparator): nasal instillation of Vardenafil ( visit 2 or 3)
  Interventions: Drug: Vardenafil
- Placebo (Placebo Comparator): Nasal instillation of placebo (visit 3 or 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil — Nasal instillation of Vardenafil
  Arms: Vardenafil
Drug: Placebo — Nasal instillation of placebo matching in appearance with the Vardenafil instillation
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of a nasal instillation of Vardenafil on nasal potential difference in cystic fibrosis patients homozygous for the F508del mutation

DETAILED DESCRIPTION:
CFTR protein has been shown to be an ohmic, small conductance channel regulated by cAMP intracellular levels that are balanced by degradation through cyclic nucleotide phosphodiesterases (PDE). Several families of PDEs with varying selectivities for cAMP and/or cGMP have been identified.PDE5 is highly specific for cGMP and is involved in the regulation of the intracellular concentration of cGMP in various tissues. Recently, it has been shown, in a preclinical model of transgenic mice, that pharmacological doses of sildenafil and vardenafil, two clinically approved PDE5 inhibitors, stimulate chloride transport activity of the mutant F508del-protein (Lubamba et al, 2008); this parameter has been assessed by means of the nasal potential difference (NPD). An increasing effect of sildenafil on the expression of F508del-CFTR protein (Dormer et al,2005) was originally reported in nasal epithelial cells harvested from patients with cystic fibrosis and cultured on impermeable supports, a configuration that allows interaction of drugs with the apical side of epithelia.

This study aims at investigating the effect of a single local administration of vardenafil on NPD measurements in CF patients homozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients homozygous for the F508del mutation as confirmed by a genetic test
* Aged 14 years and older
* Male and female
* FEV1 >50% of predicted normal

Exclusion Criteria:

* Acute respiratory tract infection or pulmonary exacerbation requiring antibiotic intervention within 2 weeks of visit 1
* Any condition prohibiting the correct measurement of the NPD
* Active or passive smoking
* Planned treatment or treatment with another investigational drug or therapy within 1 month prior to randomisation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cumulated changes in response to Chloride-free solution and isoproterenol (reflecting chloride transport) | Change from baseline (visit 1) and placebo to Vardenafil instillation

SECONDARY OUTCOMES:
Change in basal voltage value and in amiloride response (reflecting sodium transport) | Change from baseline (visit1) and placebo to Vardenafil instillation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick LEBECQUE, MD, PhD, Principal Investigator — Cliniques universitaires St.Luc (Université catholique de Louvain); Teresinha LEAL, MD, PhD, Principal Investigator — Cliniques universitaires St.Luc ( Université Catholique de Louvain); Anissa LEONARD, MD, Principal Investigator — Cliniques universitaires St.Luc (Université Catholique de Louvain)
Locations (1):
- Cliniques universitaires St. Luc, Brussels, Belgium

REFERENCES:
- [Result] Dormer RL, Harris CM, Clark Z, Pereira MM, Doull IJ, Norez C, Becq F, McPherson MA. Sildenafil (Viagra) corrects DeltaF508-CFTR location in nasal epithelial cells from patients with cystic fibrosis. Thorax. 2005 Jan;60(1):55-9. doi: 10.1136/thx.2003.019778. PMID 15618584
- [Result] Lubamba B, Lecourt H, Lebacq J, Lebecque P, De Jonge H, Wallemacq P, Leal T. Preclinical evidence that sildenafil and vardenafil activate chloride transport in cystic fibrosis. Am J Respir Crit Care Med. 2008 Mar 1;177(5):506-15. doi: 10.1164/rccm.200703-344OC. Epub 2007 Nov 15. PMID 18006891